CLINICAL TRIAL: NCT06716944
Title: A Feasibility Trial of Self-Acupuncture for Patients With Migraines (SAM)
Brief Title: Self-acupuncture for Migraines Feasibility Study
Acronym: SAM
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of West London (Other)
Responsible Party: Principal Investigator, Catrina Davy, Chief investigator, University of West London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAM
Record Dates: First submitted 2024-10-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Migraine
Keywords: migraine; acupuncture
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This study is not to test the device (acupunture0 but the trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-acupuncture plus usual care (Active Comparator): Participants will be taught to do self-acupuncture to manage their migraines. They can also do all the other things they normally do to manage their migraines apart from having acupuncture elsewhere.
  Interventions: Device: Acupuncture
- usual care (No Intervention): Participants can do all the other things they normally do to manage their migraines apart from having acupuncture elsewhere.

INTERVENTIONS:
Device: Acupuncture — self-acupuncture
  Arms: self-acupuncture plus usual care

SUMMARY:
Patients who have had a course of acupuncture at the Royal London Hospital for Integrated Medicine to manage their migraines, and found it effective, will be taught to do self-acupuncture. This is a feasibility study so the main aim is to test the trial design but the researchers will also explore self-acupuncture's effectiveness, acceptability and safety.

DETAILED DESCRIPTION:
Aim: The proposed study will evaluate the feasibility of teaching SA to patients with migraines in the United Kingdom National Health Service setting.

Methodology: The study will employ a pragmatic, mixed-methods, randomised, parallel-group, exploratory design. The study will compare SA plus standard care versus standard care alone. Participants will complete outcome measures at various time points and be invited to take part in a qualitative telephone interview to explore their views on the design of the study and acceptability of the intervention. The researcher will take field notes of the observation of the SA teaching session to explore the acceptability of the SA teaching method. Data will be analysed to test the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years old and over.
* Patients with migraines (when topiramate and propranolol are unsuitable).
* Patients who have been referred to the Royal London Hospital for Integrated Medicine (RLHIM) for a course of at least 6 acupuncture sessions to manage their migraines.
* Patients who have completed a course of acupuncture for the management of their migraines at RLHIM and self-declare that they benefitted from it.
* Patients must have completed the course of acupuncture within the last 3 to 24 months.

Exclusion Criteria:

* Patients unwilling to participate (for instance due to needle phobia).
* Patients currently receiving acupuncture.
* Patients with severe clotting dysfunction or who bruise spontaneously.
* Patients unable to complete the questionnaires as judged by the researchers.
* Patients who have previously been taught or have practiced SA.
* Patients who are assessed as being unable to do SA (such as if they have poor hand function).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Test (HIT6) | From enrolment to end of intervention at 24 weeks
  HIT-6 assesses the burden of headaches (including migraine) by assessing the impact of headaches on peoples' daily living, work and social situations. Patients rate six areas of potential impact on a 5-part scale from 'never' to 'always'.

OTHER OUTCOMES:
Migraine Disability Assessment (MIDAS) | From enrolment to end of intervention at 24 weeks
  MIDAS assesses the impact headaches or migraines have on peoples' daily living. Patients record the number of days in the last three months that their migraine has impacted their work, household work and social activities (there are five items in the measure).
Migraine-Specific Quality of Life Questionnaire (MSQ v2.1) | From enrolment to end of intervention at 24 weeks
  MSQ v2.1 assesses the impact of migraine on peoples' quality of life. Patients rate how often in the last four weeks their migraine has impacted various areas of daily living. The questionnaire consists of 14 questions which relate to three areas: daily activities the patient was restricted from doing, daily activities the patient was prevented from doing and impact on emotional wellbeing. Patients can rate the impact of each item on a 6-part scale from 'none of the time' to 'all of the time'.
Pain Catastrophising Scale (PCS) | From enrolment to end of intervention at 24 weeks
  The PCS measures the impact of pain on peoples' daily living. The questionnaire consists of 13 items. Patients rate the impact pain has on these items on a 5-part scale from 'not at all' to 'all of the time'.
Migraine diary | From enrolment to end of intervention at 24 weeks
  Participants will be asked to keep a diary of their migraines. They will be asked to record the frequency, duration and severity of their migraines, other symptoms they experienced (such as dizziness or nausea), any migraine or pain medication they took and any other comments.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital for Integrated Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
I'm not sure what it involves